CLINICAL TRIAL: NCT00828724
Title: An Open Label, Single Dose, Cross-over Study to Assess the Pharmacokinetic Properties of Lorcaserin in the Fed and Fasted State
Brief Title: Pharmacokinetic Properties of Lorcaserin in the Fed and Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: APD356-015
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorcaserin 10mg (Experimental)
  Interventions: Drug: Lorcaserin 10mg

INTERVENTIONS:
Drug: Lorcaserin 10mg

SUMMARY:
The purpose of this study is to evaluate the PK properties in fed and fasted men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 18 and 65 years (inclusive)
2. Able to give signed informed consent
3. BMI 27-45 kg/m2, inclusive
4. Eligible male and female subjects must agree not to participate in a conception process.
5. Considered to be in stable health in the opinion of the Investigator.

Exclusion Criteria:

1. Prior participation in any study of lorcaserin.
2. Clinically significant new illness in the 1 month before screening
3. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol
4. History of any of the following cardiovascular conditions:

   * Myocardial infarction (diagnosed by cardiac enzyme[s] and/or diagnostic ECG), CVA, TIA or RIND within 6 months of screening;
   * Cardiac arrhythmia requiring medical or surgical treatment within 6 months of screening
   * Unstable angina
   * History of pulmonary artery hypertension
5. Positive result of HIV, hepatitis B or hepatitis C screens
6. Malignancy within 2 years of the screening visit (except basal cell or squamous cell carcinoma with clean surgical margins)
7. Initiation of a new prescription medication within 1 month prior to screening.
8. Recent history (within 2 years prior to the screening visit) of alcohol or drug/solvent abuse or a positive screen for drugs of abuse at screening.
9. Participated in any clinical study with an investigational drug, biologic, or device within 1 month prior to screening
10. Use of SSRIs,SNRIs, and other medications must meet the washout period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic properties of a single oral dose of lorcaserin in the fed versus fasted state

CONTACTS AND LOCATIONS:
Locations (1):
- CRI Worldwide, Willingboro, New Jersey, United States